CLINICAL TRIAL: NCT01303393
Title: Information Needs After Surgery for Colorectal Cancer - From the Perspective of the Patient and Next of Kin
Brief Title: Information Needs After Surgery for Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Jan Johansson, MD, Associate professor, Dpt of Surgery, Lund University, Sweden
Other Study IDs: Etics review Dnr 558/2006
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Colorectal Cancer
Keywords: Patient education. Patient discharge. Needs assessment.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgery for colorectal cancer: Patients that had surgery for colorectal cancer without receiving a stoma, and their next of kin.

SUMMARY:
Aim The overall aim was to investigate information needs after surgery for colorectal cancer and factors explaining information needs, both from the patients' perspective and the next of kin's.

DETAILED DESCRIPTION:
Sample Inclusion criteria are patients over 18 years of age that have gone through a surgery for colorectal cancer without having a stoma, and their next of kin with whom they live.

Instruments In study I, 100 patients filled in four different instruments 1-2 weeks after discharge to measure: QOL, information needs, sense of coherence and performance status.

QLQ-C30 and QLQ-CR38 were used to measure QOL. INFO26 were used to measure received information. The SOC - Sense of Coherence was used to measure sense of coherence. And finally the scale for ECOG Performance Status was used to measure the level of physical performance status.

In study II the same patients filled in the same instruments a second time, 5-7 week after discharge.

Information about marital status, occupation, diagnosis and prognosis were taken from the medical record.

Interviews In study III 16 patients both filled in the instruments in study I and II, and were interviewed to gain a deeper understanding of their information needs. The interviews were semi structured and will be analysed with content analysis.

In study IV the next of kin to patients in study III were interviewed about their own information needs in connection to discharge.

The interviews were performed twice for each person, 1-2 weeks after discharge and a second time, 5-7 week after discharge.

Data sampling The data were collected consecutively, and every third patient living together with their next of kin were asked to participate in the interviews.

ELIGIBILITY:
Inclusion Criteria:

* adult over 18 years of age
* surgery for colorectal cancer in one of the three hospitals in the study
* speak and read Swedish
* be able to understand the instructions written in the questionnaires

Exclusion Criteria:

* receiving a stoma
* don't want to participate
* not completed at least half of the items in both questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria are patients over 18 years of age that have had a surgery for colorectal cancer without having a stoma, and their next of kin with whom they live. They should be able to speak and read Swedish.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

SECONDARY OUTCOMES:
Information needs - patients' and next of kins' | 7 weeks
  In the interviews with patients and next of kins separately they are asked to express their needs for information at that time.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lithner, RN, Principal Investigator — Surgical clinic, Lund, Sweden
Locations (3):
- Sweden (3):
  - Surgical clinic, Helsingborg, Skåne County
  - Surgical clinic, Lund, Skåne County
  - Surgical clinic, Malmo, Skåne County